CLINICAL TRIAL: NCT06104631
Title: A 10-week Randomized Double-blinded Crossover Trial of BiOkuris® Chitin-glucan Based Formulation Versus Placebo in Patients With Crohn's Disease in Remission and Having Irritable Bowel Syndrome-like Symptoms
Brief Title: A Prospective Trial in Patients With Crohn's Disease in Remission and Having Irritable Bowel Syndrome-like Symptoms
Acronym: Relieve
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biokuris s.a. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: BK-IBSLike-2302
Record Dates: First submitted 2023-10-17; First posted 2023-10-27 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-02

CONDITIONS: Irritable Bowel Syndrome-like Symptoms; Crohn Disease Remission
Keywords: chitin-glucan; Crohn; IBS; Irritable Bowel Syndrome-like

STUDY DESIGN:
Intervention Model Description: This is a randomised, double-blind, placebo controlled, multicentre, crossover study of BK003 in adult patients with Crohn's disease in remission without treatment or with stable maintenance therapy and having IBS-like symptoms. Patients will be recruited in the university hospitals of Liège (Belgium) and Lille (France). The recruitment period will last 1 year.
  This study will consist of a 2 to 3-week run-in period. Then, patients will take either placebo or BK003 for 4 weeks, stop for 2 to 3 weeks (washout) and then switch products for 4 additional weeks.
  Patients will undergo 5 visits: V0 (screening visit), V1 (randomization visit, 2 to 3 weeks ± 4 days after V0), V2 (washout, 4 weeks ± 4 days after V1), V3 (crossover, 18 days ± 3 days after V2) and V4 (end of study visit, 4 weeks ± 4 days after V3).
Who Masked: Participant, Investigator
Masking Description: At V1, all enrolled patients will be randomly allocated to either BK003 or placebo using computerised block-randomisation with a 1:1 ratio. The randomisation list has been generated before study product packaging and each product has a number which will be consecutively allocated to patients in the eCRF.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BK003 (Experimental): Dietary Supplement: BK003 The product is a combination of chitin-glucan and micronutrients. The dose of chitin-glucan is 3 g/day. The product is provided as sachets containing powder to be dissolved in a glass of water (about 250 ml) and taken orally.
  Interventions: Other: BK003
- Placebo (Placebo Comparator): Dietary Supplement: BK003 placebo The placebo product has the same composition in excipient, same form and same posology as BK003.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: BK003 — The product is a combination of chitin-glucan and other dietary complement components. The dosage of chitin-glucan is 3 g/day. The product is a powder for oral administration 1x/day.
  Arms: BK003
Other: Placebo — The placebo product has the same composition in excipient, same form and same posology as BK003.
  Arms: Placebo

SUMMARY:
Crohn's disease is a chronic and complex inflammatory bowel disease affecting the gastrointestinal tract, causing symptoms like abdominal pain, diarrhea, and fatigue. While its exact cause is unclear, it involves genetic, environmental, and immunological factors. Crohn's disease can lead to nutrient deficiencies and has unpredictable flare-ups and remission periods. During the remission phases, irritable bowel syndrome (IBS)-like symptoms can persist in 50% of patients, for which no satisfactory treatment is available yet.

Chitin-glucan is prebiotic, obtained by extraction, isolation and purification from a fungal resource: the mycelium of Aspergillus niger (a microscopic fungus of the Ascomycetes family) of which it composes the cell walls. The biopolymer consists essentially of two types of polysaccharide chains: chitin (poly-N-acetyl-D-glucosamine) and beta-(1,3)-D-glucan (D-glucose units linked essentially via beta-1,3 bonds). Because of its beta bond, human intestinal enzymes cannot digest it, as a result, the majority of chitin-glucan can reach the colon where it can be fermented by the microbiota.

By modulating the composition and/or activity of the intestinal microbiota, fermentation of chitin-glucan could have beneficial effects on health.

The aim of the RELIEVE study is to assess if BK003 could improve the relief of global symptoms, individual symptoms, stool consistency and frequency of evacuations, quality of life, anxiety, and depression in patients with Crohn's disease in remission without treatment or with stable maintenance therapy and having IBS-like symptoms and to confirm the product's safety.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged from 18 years to 75 years,
* Long standing (>3 months prior to V1) steroid-free clinical remission Crohn's disease according to clinical and biochemical assessments,
* Clinical remission (according to the investigator),
* Absence of inflammatory markers at V1,
* Presence of IBS-like symptoms according to Rome IV criteria,
* Likert scale ≥ 3 for abdominal pain at V0,
* Patient with correct and complete reporting of the study questionnaires and scores during the run-in period (≥ 75% completion),
* To continue all medication used in the last month before inclusion at the same dosage,
* Anti-spasmodic, hypomotility agents, probiotics, prebiotics, bile-acid chelators, and anti-depressants are authorized if consumed for longer than 1 month before inclusion and maintained at a stable dosage for the entire study duration,
* Agreeing to maintain their lifestyle behaviours during the participation in the study,
* Patient has read, understood, and signed the informed consent form (ICF),
* Patients capable of communicating with the investigator, replying to the questionnaires, and understanding the requirements and constraints of the study protocol,
* Possession of a digital device (i.e., smartphone or tablet),
* Patient willing to adhere to the study visit schedule and able to understand and comply with protocol requirements and product administration,
* Male or female patient of childbearing potential who agrees to use acceptable methods of birth control (oral, transdermal, systemic contraception, intrauterine device, condom) for the duration of the study,
* Patient can read and write in French.

Exclusion Criteria:

* Patients with other concomitant organic gastrointestinal abnormalities besides Crohn's disease: ano-perineal lesions, extra-intestinal manifestations of Crohn's disease, colorectal history of cancer or abdominal radiotherapy, symptomatic intestinal stenosis, substance dependence history,
* Patients with significant comorbidities: instable cardiovascular diseases, complicated diabetes, instable thyroid function,
* Patients receiving non-steroidal anti-inflammatory drugs, steroids, opioids, or narcotic analgesics in the last month before V0,
* Patients beginning a diet or a specific treatment for functional symptoms (probiotics, prebiotics, anti spasmodic, chelators, anti-depressants, etc.) within one month before V1,
* Ongoing antibiotics or antibiotics prescribed in the last 2 weeks before V1.
* Excessive alcohol consumption (>30 g/day [i.e., 3 units/day] for men and >20 g/day [i.e., 2 units/day] for women) and/or drug abuse,
* Pregnancy and lactation, or plan to become pregnant during the study period,
* Participation in other studies involving investigational or marketed products concomitantly or less than 3 months prior to V0,
* Known hypersensitivity to any of the ingredients or excipients of the study products,
* Patient who has forfeited their freedom by administrative or legal award, or who is under guardianship or under limited judicial protection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Subject's global assessment (SGA) | at week 4 after randomization on period I (cross over) and at week 4 after wash-out period II (cross over)
  Subjective global assessment of relief responder rate. SGA is scored on a 5-point Likert scale (1 = completely relieve and 5= being worse). Patients with an SGA of relief score from 1 to 3 is considered as responder.

SECONDARY OUTCOMES:
Individual symptoms | weekly from randomization up to the end of the study (week 10 post run in)
  Weekly change from baseline in mean 7-point Likert scale for each of the symptoms: abdominal pain, abdominal bloating, flatulence. Scores of each symptoms will be assessed (from 1= none to 7= very severe) every day and mean scores of each symptoms will be calculated every week of the treatment period I & II and compared with baseline (run-in period).
Stool consistency & dyschesia | weekly from randomization up to the end of the study (week 10 post run in)
  Weekly change from baseline on number of normal stool. BSS score, including dyschesia, will be assessed every day and mean scores will be calculated every week until the end of the study
Stool number | weekly from randomization up to the end of the study (week 10 post run in period)
  Weekly change from baseline on number of evacuations per day. The mean daily number of bowel movements will be calculated for each week until the end of the study
IBS-related quality of life | At week 0, week 4, week 6, week 10 post-run in period
  The absolute and relative change of IBS-related quality of life score.
Anxiety and depression | At week 0, week 4, week 6, week 10 post-run in period
  The absolute and relative change of anxiety and depression (HADS score)
Serum CRp & fecal calprotectine | at week 4 versus week 0 (period I) and at week 10 versus week 6 (period II) post run in period
  Change from baseline for the following measures : serum CRP, fecal calprotectine, alpha diversity and the relative abundance of bacterial, viral and fungal taxa in stools
Adverse events | At week 0, week 4, week 6, week 10 post-run in period
  Occurence and severity of adverse events

CONTACTS AND LOCATIONS:
Locations (2):
- CHU Liege - Gastroenterology, Liège, Belgium
- CHU Lille - Gastroenterology, Lille, France